CLINICAL TRIAL: NCT07323199
Title: High-Intensity Interval Training (HIIT) and Transcranial Direct Current Stimulation (tDCS) in Women With Fibromyalgia - Effects on Clinical and Neuro-physiological Variables: Randomized Clinical Trial Protocol
Brief Title: Exercise and Neuromodulation in Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Edith Elgueta Cancino, Associate Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33B2024
Record Dates: First submitted 2025-09-30; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia (FM)
Keywords: Fibromyalgia; central sensitization; Pain; intracortical excitability; HIIT - HIGH-INTENSITY INTERVAL TRAINING; tDCS - transcranial direct stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Exercise; Dosage Forms; Neurotransmitter Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants from tDCS (active) and sham tDCS (inactive) groups will be blinded to the stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIGH-INTENSITY INTERVAL TRAINING (HIIT) plus active TRANSCRANIAL DIRECT CURRENT STIMULATION (tDCS) (Experimental): The participants will cycle with a HIGH-INTENSITY INTERVAL TRAINING protocol while being stimulated with active TRANSCRANIAL DIRECT CURRENT STIMULATION for 20 minutes. This intervention will be performed three times per week for four weeks.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION; Other: Neuromodulators
- HIGH-INTENSITY INTERVAL TRAINING (HIIT) plus sham TRANSCRANIAL DIRECT CURRENT STIMULATION (tDCS) (Sham Comparator): The participants will cycle with a HIGH-INTENSITY INTERVAL TRAINING protocol while being stimulated with sham TRANSCRANIAL DIRECT CURRENT STIMULATION for 20 minutes.
  During exercise intervention, to replicate the feeling of current ramping up during active stimulation, the active anode placed on the left M1 will be activated for 30 seconds at the beginning and end of the procedure.
  This intervention will be performed three times per week for four weeks.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION; Other: Neuromodulators
- HIGH-INTENSITY INTERVAL TRAINING (HIIT) (Active Comparator): The participants will cycle with a HIGH-INTENSITY INTERVAL TRAINING protocol for 20 minutes without any stimulation.
  This intervention will be performed three times per week for four weeks.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — HIIT training: The participants will perform a HIIT protocol that consists of 1 minute of cycling at 50-60 revolutions per minute with a load that generates an effort of 80%-95% of their maximum Heart Rate (HR). Then 2 minutes of passive recovery, all this repeated 10 times (1x2x10). The effort of the session will be monitored by rating the perceived exertion (RPE) with a scale from 6-20 and HR. If the participant fails to recover within 2 minutes (>70% maximum heart rate), resting time will be extended until an HR ≤ 70% of the maximum is achieved. The maximum HR of each session will be used for HIIT prescription for the next session.
Other: Neuromodulators — Active tDCS: Two electrodes covered by a damp sponge will be placed on the scalp. The active electrode (anode) will be placed on the left motor cortex and the cathode on the contralateral supraorbital area before the exercise starts. The stimulation will start at the same time as the exercise, with an intensity of 2mA for 20 minutes.
  Arms: HIGH-INTENSITY INTERVAL TRAINING (HIIT) plus active TRANSCRANIAL DIRECT CURRENT STIMULATION (tDCS); HIGH-INTENSITY INTERVAL TRAINING (HIIT) plus sham TRANSCRANIAL DIRECT CURRENT STIMULATION (tDCS)

SUMMARY:
Exercise is recommended for people with fibromyalgia because it can reduce symptoms and improve quality of life. Some studies show that high-intensity exercises like running or cycling (also called high-intensity interval training, or HIIT) may reduce symptoms more effectively than slower, traditional exercises.

There are also new treatments, like non-invasive neuromodulation, which uses a gentle current to stimulate brain cells. This technique can help reduce pain in people with fibromyalgia. However, we don't yet know if combining HIIT and neuromodulation works better than exercise alone. We also want to find out if this combination helps improve other symptoms like fatigue and poor sleep.

The goal of this study is to see how a combination of HIIT and neuromodulation affects pain, fatigue, sleep, and muscle strength in women with fibromyalgia.

The investigators are asking two main questions:

Does combining HIIT and neuromodulation reduce pain better than exercise alone? Does this combination improve how the brain controls pain, muscles, and other symptoms like fatigue and sleep problems? What Will the Study Involve?

Three different exercise training programs will be compared:

HIIT with neuromodulation (tDCS): The participant will do HIIT by cycling at a high intensity for 1 minute, then resting for 2 minutes. Then, this will be repeated 10 times. At the same time, the researchers will place two small, damp sponges on the head of the participant. These sponges connect to the tDCS device, which sends a gentle current to your brain. It might feel a tingling sensation at first, but it will fade away.

HIIT with a "sham" (inactive) neuromodulation: This is similar to the first program, but the tDCS device will only be active for a few minutes at the beginning and end of the session.

HIIT alone: This involves just the cycling exercise with no brain stimulation. Who Can Participate?

The researchers are looking for women who:

Are 18-65 years old and have been diagnosed with fibromyalgia Experience moderate to high levels of pain Have stable blood pressure (if they have hypertension) Are not regularly active (don't do more than 30 minutes of exercise at least 3 times per week)

What Will the Study involve?

The participant will:

Attend 6 conditioning sessions (cycling) over two weeks to prepare their body. Complete 4 weeks of HIIT training, three times per week, at Universidad Andres Bello.

Attend 3 assessment sessions in our lab: before the conditioning, before the training, and after the training. These will include:

Non-invasive tests to measure your physical fitness, muscle strength, and pain sensitivity Brain and muscle connection tests. Questionnaires about your sleep, pain, fatigue, anxiety, depression, and exercise enjoyment

What the participant will get?

At the end of the study in addition to the training benefits, participants will receive a detailed report showing their body composition (muscle and fat levels) before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of Fibromyalgia by a physician according to the criteria of the American College of Rheumatology (ACR) 2016
* A stable medical treatment for symptoms for at least 4 weeks before participation (stable doses of medication)
* Reported pain equal to or higher than 40 mm on the visual analogue scale (moderate or severe pain) for more than 3 months
* Body mass index (BMI) between 18.5 and 39.9 kg m-2,
* Controlled high blood pressure.

Exclusion Criteria:

* Isolated inflammatory joint, cancer, infectious, traumatic, localised neuropathic or degenerative joint pain.
* Intense headache, cerebral surgery, seizure/epilepsy, cardiovascular, lung, metabolic (II diabetes mellitus), retinopathy or neurological diseases (i.e. stroke and traumatic brain injury antecedents),
* Severe psychiatric disorders, major depression
* Substance abuse.
* Currently pregnant/breastfeeding,
* Under physical therapy treatment or have participated in a designed sports or exercise training in systematic programs in the last 3 months.
* Unable to speak or read Spanish fluently (inability to understand the pain scale and cooperate in testing)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Changes of the numeric rating scale (0-10) for pain severity | Participants will be asked to rate their pain sensation at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The primary outcome is the auto reported rating of pain severity with a numeric rating scale from 0 to 10 points. Commonly used to assess pain severity, where zero means "no pain" and 10 means "the worst pain imaginable". Participants will be asked to rate their pain sensation before and after the intervention.

SECONDARY OUTCOMES:
Changes in generalised perception of fatigue | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Generalised Fatigue: "is a profound and overwhelming, more severe, constant, and unpredictable than normal tiredness, not relieved by resting or sleep, not proportional to effort exerted, and disruptive in terms of motivation, activities, and cognition". The generalised fatigue will be assessed with:
  Multidimensional Fatigue Inventory (MFI). A questionnaire with 20 items divided into 5 domains: general fatigue, physical fatigue, mental fatigue, reduced activity and reduced motivation. The score range is between 4 to 20 points; a higher score indicates a greater degree of fatigue.
Changes in generalised perception of fatigue | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The Symptom Severity (SS) Score, a tool that measures the severity of symptoms like fatigue, unrefreshed sleep, and cognitive issues, along with other somatic symptoms, over the past week. Rating the severity from 0 (no problem) to 3 (severe).
Changes in generalised perception of fatigue | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Fibromyalgia Impact Questionnaire (FIQR): The sub-item evaluates fatigue with a rating scale of 11 blocks (0 to 10). Higher scores indicate no energy.
Changes in sleep quality | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The sleep quality will be measured with:
  Numeric Rating Scale (0-10): single-item tool that instructs the patient to describe the quality of sleep during the past 24 hours, where 0 is the best possible sleep and 10 is the worst possible sleep.
Changes in sleep quality | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The sleep quality will be measured with:
  Pittsburgh Sleep Quality Index (PSQI): a questionnaire that assesses duration, disturbance, latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality and sleep medication use. Each component is scored from 0 to 3. Low scores indicate good sleep quality and high scores indicate poor sleep quality. (0-4: Good sleep quality; 5-10: Poor sleep quality; >10: Very poor sleep quality).
Changes in the level of depression | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Depression will be assessed with two the subitem for depression of the "Fibromyalgia Impact Questionnaire (FIQR)". This goes from 0 to 10 in an 11-point rating scale with higher scores representing severity.
Changes in the level of depression | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Beck's Depression Inventory II (BDI-II): a 21-item self-reported measure that assesses the cognitive, affective, and neurovegetative symptoms of depression. The total score is 63 points. The range score is 0-13 "minimal", 14-19 "mild", 20-28 "moderate" and 29-63 "severe".
Changes in quality of life | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Quality of life will be assessed with the "Fibromyalgia Impact Questionnaire (FIQR)", which is a 21-item self-administered questionnaire. The questionnaire has 3 domains: function, overall impact and symptoms. The total score ranges from 0 to 100 points; higher scores indicate a severe impact.
Changes in quality of life | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Quality of life will be assessed with the "Short Form-36 (SF-36)". This questionnaire surveys health status, assesses physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. The highest score is 100, and the higher the score, the better the quality of life.
Changes corticospinal excitability | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  To estimate corticospinal excitability peak-to-peak amplitude of the Motor Evoked Potential (MEP) will be measured. MEP is the response of the muscle to the stimulation of the corticomotor pathway with a magnetic stimulator and is measured with electromyography in milliAmpere (mA).
Adherence to training | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The adherence to exercise will be measured by the "Exercise Attitude Questionnaire". The score is 1 point "strongly disagree", 2 points "somewhat disagree", 3 points "somewhat agree", 4 points "strongly agree". The total score is 72 points, and the cut-off point for adherence is >60 points
Physical Activity | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Physical Activity Readiness Questionnaire (PAR-Q): pre-participation screening tool for detection of possible health and cardiovascular problems. Include seven health-related questions to be answered yes or no. If the answer is "yes" to one question, the participant should talk to a physician before starting physical activity. If all questions are yes, the participant is fit to perform physical activity.
Physical Activity | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  International Physical Activity Questionnaire (IPAQ): estimates the level of physical activity in different activity domains such as occupational, transport, yard/garden, household, leisure, and sitting. 27 items give a detailed picture of activity in different domains (work, transport, domestic, leisure). Measures frequency (days/week) and duration (minutes/day) of physical activity in the last 7 days, across intensity levels. It expresses activity in Metabolic Equivalent of Task (MET)-minutes per week (MET-min/week) or the energy cost of physical activities, where 1 MET is the energy expended at rest ≈ 3.5 mL O₂/kg/min. Higher values indicate greater physical activity level.
Maximal voluntary isometric contraction | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  It is the maximal voluntary effort of isometric contraction. The strength of the quadriceps will be evaluated during 3 trials using an isokinetic dynamometer (Isoforce®).
Muscle endurance | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  A knee extension at 20% maximal voluntary contraction will be performed until exhaustion. Participants' perception of effort will be measured using the 15-point rating of perceived exertion (RPE) scale every 20 seconds of the time to exhaustion task.
Aerobic capacity | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The aerobic capacity will be measured during an incremental cycling test. During this test, will be determined the maximum oxygen consumption (VO2peak) and the production of maximum concentric power (POmax)
Pain Sensitivity | Participants will be asked to rate their pain sensation at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Pressure will be applied at an increasing rate of 50 kPa per second with an algometer placed perpendicular over the skin until the sensation of pressure changes to pain also known as pain pressure threshold (PPT).
Muscle soreness | Participants will be asked to rate their pain sensation at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  To quantify the muscle soreness, the participants must mark with a straight vertical line on the horizontal line (from 0 to 100 millimetres), after performing a task of sitting and standing 3 times.
Changes in the number of painful areas in the body | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The participant will report the number of painful areas of the body (upper, lower, or axial regions) over the last week. The total score is 19, where 1 region pain equals 1 point, divided by the left upper region, right upper region, axial region, left lower region and right lower region.
Changes in Active Motor Threshold | Participants will be assessed before (T0) and after (T1) the four-week intervention.
  It is the lowest stimulus intensity of a transcranial magnetic stimulator to generate a motor evoked potential with a peak-to-peak amplitude of 200 microvolts in at least five out of 10 consecutive trials when the muscle is activated at 20% of the maximal voluntary contraction.
Changes in Resting Motor Threshold | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  It is the lowest stimulus intensity of a transcranial magnetic stimulator to generate a motor evoked potential with a peak-to-peak amplitude of 50 microvolts in at least five out of 10 consecutive trials when the muscle is at rest.
Changes in the silence period after the motor evoked potential | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  It is the temporary interruption of the electromyographic signal from a muscle following a motor evoked potential. It is considered a measure of the excitability mediated by gamma-aminobutyric acid receptors. It will be measured in milliseconds (ms) from the end of the motor evoked potential wave to the recovery of the signal to the basal averaged amplitude.
Changes in anxiety levels | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  Changes in anxiety will be assessed with the subitem that evaluates anxiety of the "Fibromyalgia Impact Questionnaire (FIQR)" with 11 blocks (0 to 10), where higher scores indicate a severe impact.
Changes in anxiety levels | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  State Trait Anxiety Inventory (STAI) will be used to assess anxiety levels. The total score is 80 points. The score is classified as 20-37 "no or low anxiety", 38-44 "moderate anxiety" and 45-80 "high anxiety".
Level of enjoyment of exercise | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The enjoyment of exercise will be assessed with the "Physical Activity Enjoyment Scale". This scale includes 16 items with a maximum score of 80 points. The rating scale ranges from 1 ("dislike a lot") to 5 ("enjoy a lot").
Level of muscle soreness | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The participants will be asked to sit and stand 3 times with their legs shoulder-width apart and bend their knees to 90°. The volunteer must rate the level of discomfort by marking a straight vertical line on the horizontal line of a 100 mm rating scale. Higher values indicate greater soreness.
Level of fear of movement | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The fear of movement will be assessed with the Tampa Scale for Kinesiophobia. A questionnaire of 17 questions, with a maximum of 68 points. Scores > 37 points indicate high levels of kinesiophobia, and ˂ 37 points indicate low levels.
Changes in negative cognitions related to pain | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The catastrophization of pain will be assessed with a self-reported questionnaire designed to assess catastrophic thinking related to pain among adults. This "Pain Catastrophizing Scale" has 13 items, each describing a thought or feeling about pain. Each item is rated on a 5-point Likert scale from 0 to 4, with a maximal score of 52. Higher scores indicate high catastrophising.
Changes in negative cognitions related to pain | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The acceptance of chronic Pain will be assessed with a 20-item questionnaire, "Chronic Pain Acceptance Questionnaire for Fibromyalgia", scored with a 7-point Likert scale (0 = "never true" to 6 = "always true"). Higher scores indicate better adjustment and functioning.
Changes in body composition | Participants will be assessed at baseline, pre-intervention(T0) and immediately after the four-week intervention (T1).
  The weight and body composition in percentage of muscle, fat and water will be measured with a bioimpedanciometer (InBody 770).

CONTACTS AND LOCATIONS:
Locations (1):
- Excercise and Rehabilitation Sciences Institute, Universidad Nacional Andres Bello, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. The main reasons are related to the protection of participant confidentiality and the absence of formal mechanisms or resources to support secure data sharing. A summary of the results of the study will be published in peer-reviewed journals and presented at scientific meetings, ensuring transparency and dissemination of findings without compromising participant privacy.

REFERENCES:
- [Background] Kolak E, Ardic F, Findikoglu G. Effects of different types of exercises on pain, quality of life, depression, and body composition in women with fibromyalgia: A three-arm, parallel-group, randomized trial. Arch Rheumatol. 2022 May 7;37(3):444-455. doi: 10.46497/ArchRheumatol.2022.9190. eCollection 2022 Sep. PMID 36589612
- [Background] Angius L, Pageaux B, Hopker J, Marcora SM, Mauger AR. Transcranial direct current stimulation improves isometric time to exhaustion of the knee extensors. Neuroscience. 2016 Dec 17;339:363-375. doi: 10.1016/j.neuroscience.2016.10.028. Epub 2016 Oct 14. PMID 27751960
- [Background] Martinez-Valdes E, Falla D, Negro F, Mayer F, Farina D. Differential Motor Unit Changes after Endurance or High-Intensity Interval Training. Med Sci Sports Exerc. 2017 Jun;49(6):1126-1136. doi: 10.1249/MSS.0000000000001209. PMID 28121801
- [Background] Hooten WM, Smith JM, Eldrige JS, Olsen DA, Mauck WD, Moeschler SM. Pain severity is associated with muscle strength and peak oxygen uptake in adults with fibromyalgia. J Pain Res. 2014 May 3;7:237-42. doi: 10.2147/JPR.S61312. eCollection 2014. PMID 24833914
- [Background] Kosek E, Ekholm J, Nordemar R. A comparison of pressure pain thresholds in different tissues and body regions. Long-term reliability of pressure algometry in healthy volunteers. Scand J Rehabil Med. 1993 Sep;25(3):117-24. PMID 8248762
- [Background] Ziemann U, Lonnecker S, Steinhoff BJ, Paulus W. Effects of antiepileptic drugs on motor cortex excitability in humans: a transcranial magnetic stimulation study. Ann Neurol. 1996 Sep;40(3):367-78. doi: 10.1002/ana.410400306. PMID 8797526
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Background] Groppa S, Oliviero A, Eisen A, Quartarone A, Cohen LG, Mall V, Kaelin-Lang A, Mima T, Rossi S, Thickbroom GW, Rossini PM, Ziemann U, Valls-Sole J, Siebner HR. A practical guide to diagnostic transcranial magnetic stimulation: report of an IFCN committee. Clin Neurophysiol. 2012 May;123(5):858-82. doi: 10.1016/j.clinph.2012.01.010. Epub 2012 Feb 19. PMID 22349304
- [Background] Pacheco-Barrios K, Lima D, Pimenta D, Slawka E, Navarro-Flores A, Parente J, Rebello-Sanchez I, Cardenas-Rojas A, Gonzalez-Mego P, Castelo-Branco L, Fregni F. Motor cortex inhibition as a fibromyalgia biomarker: a meta-analysis of transcranial magnetic stimulation studies. Brain Netw Modul. 2022 Apr-Jun;1(2):88-101. doi: 10.4103/2773-2398.348254. Epub 2022 Jun 29. PMID 35845034
- [Background] Hupfeld KE, Swanson CW, Fling BW, Seidler RD. TMS-induced silent periods: A review of methods and call for consistency. J Neurosci Methods. 2020 Dec 1;346:108950. doi: 10.1016/j.jneumeth.2020.108950. Epub 2020 Sep 22. PMID 32971133
- [Background] Zeugin D, Ionta S. Anatomo-Functional Origins of the Cortical Silent Period: Spotlight on the Basal Ganglia. Brain Sci. 2021 May 27;11(6):705. doi: 10.3390/brainsci11060705. PMID 34071742
- [Background] Hoeger Bement MK, Weyer AD, Yoon T, Hunter SK. Corticomotor excitability during a noxious stimulus before and after exercise in women with fibromyalgia. J Clin Neurophysiol. 2014 Feb;31(1):94-8. doi: 10.1097/WNP.0000000000000025. PMID 24492452
- [Background] Ridding MC, Taylor JL. Mechanisms of motor-evoked potential facilitation following prolonged dual peripheral and central stimulation in humans. J Physiol. 2001 Dec 1;537(Pt 2):623-31. doi: 10.1111/j.1469-7793.2001.00623.x. PMID 11731592
- [Background] McManus WF, Walker EE, Musselman MM. Effect of hydrocortisone on the localization of endotoxin in the peripheral vascular system as determined by fluorescent antibody technique. Surg Forum. 1965;16:7-9. No abstract available. PMID 5319693
- [Background] Arturi P, Schneeberger EE, Sommerfleck F, Buschiazzo E, Ledesma C, Maldonado Cocco JA, Citera G. Adherence to treatment in patients with ankylosing spondylitis. Clin Rheumatol. 2013 Jul;32(7):1007-15. doi: 10.1007/s10067-013-2221-7. Epub 2013 Mar 21. PMID 23515597
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Rivera J, Gonzalez T. The Fibromyalgia Impact Questionnaire: a validated Spanish version to assess the health status in women with fibromyalgia. Clin Exp Rheumatol. 2004 Sep-Oct;22(5):554-60. PMID 15485007
- [Background] Salgueiro M, Garcia-Leiva JM, Ballesteros J, Hidalgo J, Molina R, Calandre EP. Validation of a Spanish version of the Revised Fibromyalgia Impact Questionnaire (FIQR). Health Qual Life Outcomes. 2013 Aug 1;11:132. doi: 10.1186/1477-7525-11-132. PMID 23915386
- [Background] Sanz J, Perdigón A, Vázquez C. The Spanish adaptation of Beck's Depression Inventory-II (BDI-II): 2. Psychometric properties in the general population. Clínica y Salud 2003;14(3):249-80.
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Background] Burwinkle T, Robinson JP, Turk DC. Fear of movement: factor structure of the tampa scale of kinesiophobia in patients with fibromyalgia syndrome. J Pain. 2005 Jun;6(6):384-91. doi: 10.1016/j.jpain.2005.01.355. PMID 15943960
- [Background] Roelofs J, Goubert L, Peters ML, Vlaeyen JW, Crombez G. The Tampa Scale for Kinesiophobia: further examination of psychometric properties in patients with chronic low back pain and fibromyalgia. Eur J Pain. 2004 Oct;8(5):495-502. doi: 10.1016/j.ejpain.2003.11.016. PMID 15324781
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Hita-Contreras F, Martinez-Lopez E, Latorre-Roman PA, Garrido F, Santos MA, Martinez-Amat A. Reliability and validity of the Spanish version of the Pittsburgh Sleep Quality Index (PSQI) in patients with fibromyalgia. Rheumatol Int. 2014 Jul;34(7):929-36. doi: 10.1007/s00296-014-2960-z. Epub 2014 Feb 8. PMID 24509897
- [Background] Martin S, Chandran A, Zografos L, Zlateva G. Evaluation of the impact of fibromyalgia on patients' sleep and the content validity of two sleep scales. Health Qual Life Outcomes. 2009 Jul 10;7:64. doi: 10.1186/1477-7525-7-64. PMID 19591683
- [Background] Munguia-Izquierdo D, Segura-Jimenez V, Camiletti-Moiron D, Pulido-Martos M, Alvarez-Gallardo IC, Romero A, Aparicio VA, Carbonell-Baeza A, Delgado-Fernandez M. Multidimensional Fatigue Inventory: Spanish adaptation and psychometric properties for fibromyalgia patients. The Al-Andalus study. Clin Exp Rheumatol. 2012 Nov-Dec;30(6 Suppl 74):94-102. Epub 2012 Dec 14. PMID 23261007
- [Background] Castelo-Branco L, Uygur Kucukseymen E, Duarte D, El-Hagrassy MM, Bonin Pinto C, Gunduz ME, Cardenas-Rojas A, Pacheco-Barrios K, Yang Y, Gonzalez-Mego P, Estudillo-Guerra A, Candido-Santos L, Mesia-Toledo I, Rafferty H, Caumo W, Fregni F. Optimised transcranial direct current stimulation (tDCS) for fibromyalgia-targeting the endogenous pain control system: a randomised, double-blind, factorial clinical trial protocol. BMJ Open. 2019 Oct 30;9(10):e032710. doi: 10.1136/bmjopen-2019-032710. PMID 31672712
- [Background] Taylor JL, Holland DJ, Spathis JG, Beetham KS, Wisloff U, Keating SE, Coombes JS. Guidelines for the delivery and monitoring of high intensity interval training in clinical populations. Prog Cardiovasc Dis. 2019 Mar-Apr;62(2):140-146. doi: 10.1016/j.pcad.2019.01.004. Epub 2019 Jan 24. PMID 30685470
- [Background] Couto N, Monteiro D, Cid L, Bento T. Effect of different types of exercise in adult subjects with fibromyalgia: a systematic review and meta-analysis of randomised clinical trials. Sci Rep. 2022 Jun 20;12(1):10391. doi: 10.1038/s41598-022-14213-x. PMID 35725780
- [Background] Hou WH, Wang TY, Kang JH. The effects of add-on non-invasive brain stimulation in fibromyalgia: a meta-analysis and meta-regression of randomized controlled trials. Rheumatology (Oxford). 2016 Aug;55(8):1507-17. doi: 10.1093/rheumatology/kew205. Epub 2016 May 5. PMID 27150193
- [Background] Teixeira PEP, Pacheco-Barrios K, Branco LC, de Melo PS, Marduy A, Caumo W, Papatheodorou S, Keysor J, Fregni F. The Analgesic Effect of Transcranial Direct Current Stimulation in Fibromyalgia: A Systematic Review, Meta-Analysis, and Meta-Regression of Potential Influencers of Clinical Effect. Neuromodulation. 2023 Jun;26(4):715-727. doi: 10.1016/j.neurom.2022.10.044. Epub 2022 Nov 23. PMID 36435660
- [Background] Atan T, Karavelioglu Y. Effectiveness of High-Intensity Interval Training vs Moderate-Intensity Continuous Training in Patients With Fibromyalgia: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1865-1876. doi: 10.1016/j.apmr.2020.05.022. Epub 2020 Jun 22. PMID 32585169
- [Background] Cogiamanian F, Marceglia S, Ardolino G, Barbieri S, Priori A. Improved isometric force endurance after transcranial direct current stimulation over the human motor cortical areas. Eur J Neurosci. 2007 Jul;26(1):242-9. doi: 10.1111/j.1460-9568.2007.05633.x. PMID 17614951
- [Background] Mendonca ME, Simis M, Grecco LC, Battistella LR, Baptista AF, Fregni F. Transcranial Direct Current Stimulation Combined with Aerobic Exercise to Optimize Analgesic Responses in Fibromyalgia: A Randomized Placebo-Controlled Clinical Trial. Front Hum Neurosci. 2016 Mar 10;10:68. doi: 10.3389/fnhum.2016.00068. eCollection 2016. PMID 27014012
- [Background] Hendy AM, Andrushko JW, Della Gatta PA, Teo WP. Acute Effects of High-Intensity Aerobic Exercise on Motor Cortical Excitability and Inhibition in Sedentary Adults. Front Psychol. 2022 Mar 17;13:814633. doi: 10.3389/fpsyg.2022.814633. eCollection 2022. PMID 35369205
- [Background] Thum JS, Parsons G, Whittle T, Astorino TA. High-Intensity Interval Training Elicits Higher Enjoyment than Moderate Intensity Continuous Exercise. PLoS One. 2017 Jan 11;12(1):e0166299. doi: 10.1371/journal.pone.0166299. eCollection 2017. PMID 28076352
- [Background] Saanijoki T, Tuominen L, Tuulari JJ, Nummenmaa L, Arponen E, Kalliokoski K, Hirvonen J. Opioid Release after High-Intensity Interval Training in Healthy Human Subjects. Neuropsychopharmacology. 2018 Jan;43(2):246-254. doi: 10.1038/npp.2017.148. Epub 2017 Jul 19. PMID 28722022
- [Background] Bodere C, Cabon M, Woda A, Giroux-Metges MA, Bodere Y, Saliou P, Quinio B, Misery L, Le Fur-Bonnabesse A. A training program for fibromyalgia management: A 5-year pilot study. SAGE Open Med. 2020 Oct 7;8:2050312120943072. doi: 10.1177/2050312120943072. eCollection 2020. PMID 33110601
- [Background] Hauser W, Klose P, Langhorst J, Moradi B, Steinbach M, Schiltenwolf M, Busch A. Efficacy of different types of aerobic exercise in fibromyalgia syndrome: a systematic review and meta-analysis of randomised controlled trials. Arthritis Res Ther. 2010;12(3):R79. doi: 10.1186/ar3002. Epub 2010 May 10. PMID 20459730
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Brosseau L, Wells GA, Tugwell P, Egan M, Wilson KG, Dubouloz CJ, Casimiro L, Robinson VA, McGowan J, Busch A, Poitras S, Moldofsky H, Harth M, Finestone HM, Nielson W, Haines-Wangda A, Russell-Doreleyers M, Lambert K, Marshall AD, Veilleux L; Ottawa Panel Members. Ottawa Panel evidence-based clinical practice guidelines for aerobic fitness exercises in the management of fibromyalgia: part 1. Phys Ther. 2008 Jul;88(7):857-71. doi: 10.2522/ptj.20070200. Epub 2008 May 22. PMID 18497301
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Kleinman L, Mannix S, Arnold LM, Burbridge C, Howard K, McQuarrie K, Pitman V, Resnick M, Roth T, Symonds T. Assessment of sleep in patients with fibromyalgia: qualitative development of the fibromyalgia sleep diary. Health Qual Life Outcomes. 2014 Jul 14;12:111. doi: 10.1186/s12955-014-0111-6. PMID 25017455
- [Background] Rehm SE, Koroschetz J, Gockel U, Brosz M, Freynhagen R, Tolle TR, Baron R. A cross-sectional survey of 3035 patients with fibromyalgia: subgroups of patients with typical comorbidities and sensory symptom profiles. Rheumatology (Oxford). 2010 Jun;49(6):1146-52. doi: 10.1093/rheumatology/keq066. Epub 2010 Mar 17. PMID 20236955
- [Background] Queiroz LP. Worldwide epidemiology of fibromyalgia. Curr Pain Headache Rep. 2013 Aug;17(8):356. doi: 10.1007/s11916-013-0356-5. PMID 23801009
- [Background] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT07323199/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT07323199/ICF_001.pdf